CLINICAL TRIAL: NCT07173075
Title: Evaluation of the Relationship Between Muscle Mass Measured by Bioelectrical Impedance Analysis and the Risk of Hemorrhagic Events Under Direct Oral Anticoagulants in the Elderly
Acronym: SARCORRHAGED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2025 SORET; 2025-A01074-45 (Other: ANSM)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Direct Oral Anticoagulant; Hemmorhage; Elderly; Muscle Mass; Sarcopenia; Denutrition
Keywords: direct oral anticoagulant; hemmorhage; bleeding; elderly; muscle mass; sarcopenia; denutrition; impedancemetry
MeSH Terms: conditions — Sarcopenia; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (patient with hemorrhagic event) (Other): Patients over 70 years old, treated with one of the two factor Xa inhibitors used in France (Apixaban, Rivaroxaban), who experienced a hemorrhagic event leading to hospitalization.
  Interventions: Diagnostic Test: impedancemetry
- Control (patient without hemorrhagic event) (Other): Patients over 70 years old, treated with one of the two factor Xa inhibitors used in France (Apixaban, Rivaroxaban), followed in consultation or admitted to the hospitalization department, free from hemorrhagic events.
  Interventions: Diagnostic Test: impedancemetry

INTERVENTIONS:
Diagnostic Test: impedancemetry — impedancemetry by the InBody S10 device, during a visit, after stabilization of the patient's blood volume, within a limit of 7 days after inclusion
  Other Names: bio-impedancemetry

SUMMARY:
This study aims to assess whether reduced muscle mass is associated with an increased risk of bleeding in the elderly receiving direct oral anticoagulant therapy.

The researchers will compare the muscle mass of patients who experienced a hemorrhage (case) with that of patients who did not (control).

Muscle mass is a key criterion in the assessment of sarcopenia and malnutrition, two conditions frequently associated with aging. Sarcopenia is characterized by a significant loss of muscle mass and strength, while malnutrition is an alteration of nutritional status, often accompanied by sarcopenia, weight loss or a low body mass index (BMI). So at the same time, we want to compare sarcopenia and malnutrition between the two groups (case and control).

Cases and controls will benefit from a consultation during which measurements will be taken: weight, height, BMI, calf circumference, impedancemetry, etc. A blood test will be taken to measure anti-Xa activity (drug activity) and any missing analyses.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 70 years
* treated with one of the two factor Xa inhibitors used in France: Apixaban, Rivaroxaban.
* For cases : hemorrhagic event causing hospitalization
* For controls : free from hemorrhagic events.

Exclusion Criteria:

* Failure to obtain a consent form
* Patient under legal protection (guardianship, curatorship, or legal safeguard)
* Recurrent bleeding from a pre-existing lesion that has not received specific treatment. For example: unexplored gastrointestinal bleeding, cutaneous bleeding from a cancerous wound with therapeutic abstention.
* Bleeding caused by high-velocity trauma, surgery, or assault
* Contraindications to impedance measurement: pacemaker, cardiac defibrillator
* Elements that may provide erroneous impedance measurement data: bilateral limb amputation, bilateral joint replacements, dialysis.
* Unable to maintain the supine position.
* Digestive absorption disorder (celiac disease, short bowel, stoma, etc.)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | from enrollment and within a limit of 7 days after inclusion.
  Appendicular muscle mass expressed in kg is measured by an InBody S10 impedance meter (Appendix 3: InBody S10 impedance meter), during a visit, after stabilization of the patient's blood volume, within a limit of 7 days after inclusion.

SECONDARY OUTCOMES:
confirmed sarcopenia | from enrollment and within a limit of 7 days after inclusion.
  This is the combination of:
  * a "reduction in muscle strength" determined by a grip strength measurement and a Timed Chair Stand Test measurement
  * a "reduction in muscle mass", determined by the primary endpoint
malnutrition | from enrollment and within a limit of 7 days after inclusion.
  According to the High Authority of Health, the diagnosis of malnutrition requires the presence of at least one phenotypic criterion and one etiological criterion.
  The phenotypic criteria are as follows (one criterion is sufficient):
  * Weight loss ≥ 5% in 1 month or ≥ 10% in 6 months or ≥ 10% compared to usual weight before the onset of the disease;
  * BMI < 22 kg/m²;
  * Confirmed sarcopenia
  The etiological criteria are as follows (one criterion is sufficient):
  * Reduction in food intake of ≥ 50% for more than 1 week, or any reduction in intake for more than 2 weeks compared to: usual food consumption or protein-energy requirements;
  * Reduced absorption (malabsorption/maldigestion);
  * Pathological situation (with or without inflammatory syndrome): acute pathology or chronic pathology or progressive malignant pathology.
severe malnutrition | from enrollment and within a limit of 7 days after inclusion.
  According to the High Authority of Health, the criteria for severe malnutrition are as follows (one criterion is sufficient):
  * BMI < 20 kg/m²;
  * Weight loss: ≥ 10% in 1 month, or ≥ 15% in 6 months, or ≥ 15% compared to the usual weight before the onset of the disease;
  * Albumin level ≤ 30 g/L.
severity of muscle mass reduction | from enrollment and within a limit of 7 days after inclusion.
  There is no definition expressing a threshold; we will consider that the lower the variation is from the median, the greater the loss of muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: julien Soret, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France